CLINICAL TRIAL: NCT03905954
Title: The Impact of a Diagnosis of Parkinson's on Work
Status: Completed | Type: Observational
Sponsor: Oxford Brookes University (Other)
Collaborators: European Parkinson's Therapy Centre (Unknown)
Responsible Party: Principal Investigator, Dr Johnny Collett, Senior Clinical Research Fellow, Oxford Brookes University
Other Study IDs: MOReS-EPTC-EPDA
Record Dates: First submitted 2019-04-04; First posted 2019-04-08 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Parkinson Disease
Keywords: employment; work; diagnosis; early support
MeSH Terms: conditions — Parkinson Disease; Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parkinson's Diagnosis: Usual care
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Usual care — For this cross sectional survey, participants will be receiving usual care according to there health care systems

SUMMARY:
Parkinson's disease leads to loss of employment on average within less than 10 years of disease onset and has been found to be associated with an increased absence from work. This combined with hospitalisation; use of secondary health services; drug usage; and caregivers needing to give up work contributed to the costs associated with the conditions. It has been estimated that early support for working age newly diagnosed would cost the government about 1.5 million Euro in the UK but might lead to a potential cost saving of over half a billion over 5 years.

The study will explore the impact of a Parkinson diagnosis on employment. The study will be survey based and will include demographic questions: age, age at diagnosis of PD, educational level, and Nationality; questions pertaining to employment type, history, and reasons for leaving if this happened; and also general health.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of Parkinson

Exclusion Criteria:

None

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A (European) community based convenience sample. The survey will be available to the European Parkinson's Disease Association (EPDA) network using the Members' forum and website and will be sign posted through ongoing Member Outreach communication channels.
Sampling Method: Non-Probability Sample
Enrollment: 696 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-04 (Actual)

PRIMARY OUTCOMES:
Main occupation in the last 7 days | baseline only (cross sectional)
  Questions asks: 'Which of these descriptions applies to your main occupation in the last seven days? and has the following options.
  'In paid work (OR AWAY TEMPORARILY) (employee, self-employed, working for your family business) Unemployed and actively looking for a job Unemployed, wanting a job but not actively looking for a job Permanently sick or disabled In community or military service Doing housework, looking after children or other persons Retired In paid work (OR AWAY TEMPORARILY) (employee, self-employed, working for your family business) Unemployed and actively looking for a job Unemployed, wanting a job but not actively looking for a job Permanently sick or disabled In community or military service Doing housework, looking after children or other persons Retired Student

SECONDARY OUTCOMES:
Type of Work | baseline only (cross sectional)
  Questions asks: 'Which category would best describe your current main occupation or skill set?' Managers or directors Professionals Technicians and Associate Professionals Clerical Support Workers Services and Sales Workers Skilled Agricultural, Forestry, and Fishery Workers Craft and Related Trades Workers Plant and Machine Operators and Assemblers Elementary Occupations eg salespersons, domestic, helpers, porters Armed Forces Occupations
Symptom Severity-Distress | baseline only (cross sectional)
  0-10 visual analogue scale (0 worst - 10 best)
Symptom Severity-Pain | baseline only (cross sectional)
  0-10 visual analogue scale (0 worst - 10 best)
Symptom Severity-Fatigue | baseline only (cross sectional)
  0-10 visual analogue scale (0 worst - 10 best)
Symptom Severity-Depression | baseline only (cross sectional)
  0-10 visual analogue scale (0 worst - 10 best)
Symptom Severity-Anxiety | baseline only (cross sectional)
  0-10 visual analogue scale (0 worst - 10 best)
Symptom Severity - Sleep | baseline only (cross sectional)
  0-10 visual analogue scale (0 worst - 10 best)
Single Item Physical activity | baseline only (cross sectional)
  Days per week of physical activity lasting 30 minutes or longer on a 0-7 integer scale
Single Item Diet | baseline only (cross sectional)
  Portions of fruit and vegetables consume per day on a 0-5+ integer scale

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford Brookes University, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided